CLINICAL TRIAL: NCT01027403
Title: Evaluation of Circulating Levels of Adult Stem Cells in the Peripheral Blood of Patients With Acute Decompensated Heart Failure and Following Stabilization, in Comparison With Healthy Volunteers
Acronym: CIRCSTEM-HF
Status: Completed | Type: Observational
Sponsor: Monash University (Other)
Collaborators: The Alfred (Other)
Responsible Party: Principal Investigator, Prof Henry Krum, Professor, Monash University
Other Study IDs: 234/07
Record Dates: First submitted 2009-12-04; First posted 2009-12-08 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure
Keywords: Heart failure; Adult stem cells; Circulating stem cells; Acute decompensated heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy volunteers
- Acute decompensated heart failure

SUMMARY:
Despite advances in medical technology, heart failure remains a major cause of illness on a global scale. Medical research, over recent years, has shown that adult stem cells (as opposed to embryonic stem cells) are present in most organs of adult humans. Their exact function is however poorly understood. An improved understanding of what these stem cells do and how they work is essential if effective stem cell treatments are to be developed in future.

The project seeks to examine the levels of a number of different types of stem cells in patients with heart failure, compared to healthy volunteers. The project also aims to measure stem cell levels in patients with heart failure at the time of a sudden worsening in their condition and then later in the same patients following recovery.

The project entails the taking of blood samples in order to measure the stem cell levels in the blood. The study does NOT involve any form of treatment with stem cells. Two groups of patients will be studied; patients with heart failure and healthy volunteers.

DETAILED DESCRIPTION:
Despite advances in medical technology, heart failure remains a major cause of illness on a global scale. The quest for understanding this condition and developing new treatment strategies has led to the consideration of stem cells as a possible therapy. Medical research, over recent years, has shown that adult stem cells (as opposed to embryonic stem cells) are present in most organs of adult humans. Their exact function is however poorly understood. An improved understanding of what these stem cells do and how they work is essential if effective stem cell treatments are to be developed in future.

A number of stem cell research groups around the world have found that adult stem cells circulate in the blood of humans. These circulating cells are likely to have entered the bloodstream from the bone marrow and are thought to be traveling in the blood to get to other body organs where they may help repair damaged tissue. Interestingly, the levels of these circulating stem cells have been found to be different in healthy people compared to those with various diseases, including heart attacks and heart failure. This has lead researchers to think that these stem cells may play an important role in how the human body fights these diseases.

To date, levels of only one type of stem cell have been measured in patients with heart failure. Also, no one has studied stem cell levels in patients with heart failure at the time of a sudden worsening in their condition and then later in the same patients following recovery. This information would be very valuable in expanding scientific knowledge of these stem cells and how they behave in the different stages of heart disease.

The project seeks to examine the levels of a number of different types of stem cells in patients with heart failure, compared to healthy volunteers. The project also aims to measure stem cell levels in patients with heart failure at the time of a sudden worsening in their condition and then later in the same patients following recovery.

The project entails the taking of blood samples in order to measure the stem cell levels in the blood. The study does NOT involve any form of treatment with stem cells. Two groups of patients will be studied; patients with heart failure and healthy volunteers. Following the obtainment of informed consent, a screening history, physical examination and routine blood tests will be performed. After this, a 50ml sample of blood will be taken from the study participant. This is equivalent to 10 teaspoonfuls of blood. The 50ml blood sample obtained will then be taken immediately to the laboratory for analysis.

In the case of patients with heart failure, in order to measure stem cell blood levels after recovery, one additional blood sample will be obtained; a 50ml blood sample just before the patient is sent home from hospital.

Patients with heart failure will be identified by health care staff at the Alfred Hospital. Healthy volunteers will be identified by use of a database of healthy volunteers who have expressed interest in participating in clinical studies. Potential study participants will be initially approached and provided with written information. If the potential participant wishes to proceed with the study, this involves one outpatient hospital visit for healthy volunteers. For patients with heart failure, the study involves two visits by study staff during the hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years or older
* Hospitalized for the management of ADHF or diagnosed with ADHF within 48 hours after being hospitalized for another reason (patients/cases ONLY)
* Signed (by the subjects or their legally acceptable representatives) informed consent

Exclusion Criteria:

* Hospitalized for > 48 hours before study enrollment
* Likely to be discharged from the hospital in 24 hours or less
* Current haematological disorder or haematological malignancy
* Active infection / sepsis
* Major organ insufficiency (other than heart failure in heart failure patients)
* Pregnancy
* Healthy volunteers found to have signs and/or symptoms of heart failure on screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute decompensated heart failure and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in circulating levels of adult stem cells in the peripheral blood of patients with acute decompensated heart failure and following stabilization, in comparison with healthy volunteers. | Baseline and following stablization of heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS FRACP PhD, Principal Investigator — Monash University / Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia